CLINICAL TRIAL: NCT04094051
Title: A Retrospective and Prospective Observational Study of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) Treatment and Ibrutinib Treatment of CLL/SLL in Routine Clinical Practice
Brief Title: Observational Study of CLL/SLL Treatment and Ibrutinib Treatment of CLL/SLL in Routine Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JNJ-54179060
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ibrutinib — In the retrospective period, clinical information of approximate 500 patients with CLL/SLL prior to the study initiation will be collected retrospectively through chart review. There will be one time follow-up to collect data on disease progression, survival status and patient-reported outcomes.

SUMMARY:
This is a non-interventional, Phase 4 study designed to improve understanding of current clinical practice in the treatment of CLL/SLL and to describe treatment pattern and evaluate outcomes of ibrutinib-treated CLL patients in China. This study will include both retrospective and prospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* In the retrospective part:

  1. Male or female patients above 18 years old
  2. Patients underwent CLL treatment after Jan 1st, 2013
  3. Patient understand and voluntarily sign an ICF, if applicable.
* In the prospective part:

  1. Male or female patients above 18 years old
  2. Patients diagnosed with CLL，including treatment- naïve patients or patients who have received ≤3 prior therapies
  3. Patients treated with ibrutinib as monotherapy or a part of combination therapy
  4. Patient understand and voluntarily sign an ICF.

Exclusion Criteria:

* In the retrospective part:

  1. Patients with documented diagnosis of other cancers prior to the diagnosis of CLL
  2. Patients enrolled in interventional clinical trials of any drug for CLL treatment
* In the prospective part:

  1. Patients with documented diagnosis of other cancers prior to the diagnosis of CLL
  2. Patients with contraindication listed in the package insert of ibrutinib
  3. Patients enrolled in interventional clinical trials of ibrutinib or any other drug for CLL treatment
  4. Patient received Ibrutinib treatment as maintenance therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective group: CLL/SLL patients who received CLL/SLL treatment before study initiation as judged by participating site physician. A telephone follow-up will be arranged at the time of study initiation to determine the disease progression, survival status, PRO assessments and ADR. If the patient is accessible, oral consent will be obtained and documented in the medical record before the retrospective data collection through chart review. If the patient is not accessible at the time of study initiation, ICF waiver approved by the IRB will be in place for the etrospective data collection according to the latest local regulation. Prospective group: CLL/SLL patients who are on ibrutinib treatment at the time of study initiation as judged by participating site physician or start ibrutinib treatment after study initiation. This group of patients can be divided into two subgroups.
Sampling Method: Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient and disease characteristics | Up to 10 years
  age, gender, Eastern Cooperative Oncology Group (ECOG), stage, Bulky disease, Cytogenetics, median ANC, median hemoglobin, median platelets, comorbidity.
Treatment pattern | Baseline
  number of prior therapies, every treatment regimen, dose, cycle/treatment duration, stem cell therapy (SCT), progression-free survival (PFS), overall survival (OS), patient-reported outcome.

SECONDARY OUTCOMES:
Treatment response | Up to 10 years
  PFS, ORR, OS, minimal residual disease(MRD), patient-reported outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China